CLINICAL TRIAL: NCT05035615
Title: Evaluation of the BD OneFlow Acute Leukemia Panel (BD OneFlow ALOT, BCP-ALL T1, and AML T1-T4) on the BD FACSLyric Flow Cytometer Using Leftover, De-identified Specimens
Brief Title: Evaluation of the BD OneFlow Acute Leukemia Panel on the BD FACSLyric Flow Cytometer
Status: Completed | Type: Observational
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CAS-OFLYRICALL-IVDR
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-10

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Remnant/ Leftover specimens: Specimens that meet inclusion/exclusions criteria, are leftover from routine flow cytometry testing, and are from subjects having or suspected of having a hematological or non-hematological disorder.
  Interventions: Diagnostic Test: IUO Acute Leukemia Panel

INTERVENTIONS:
Diagnostic Test: IUO Acute Leukemia Panel — This Investigational Panel , comprised of 6 reagents , is intended for in vitro diagnostic use for qualitative flow-cytometric immunophenotyping of immature hematopoietic cell populations. These reagents are used as an aid in the differential diagnosis of hematologically abnormal patients having, or suspected of having, B-cell acute lymphoblastic leukemia or acute myeloid leukemia.

SUMMARY:
This study is a multi-site, prospective performance study to determine equivalency between the investigational OneFlow Acute Leukemia Panel on the FACSLyric system versus the final clinical diagnosis.

DETAILED DESCRIPTION:
Hematology laboratories rely on flow cytometry technology (in addition to classic hematological methods) to aid in screening, diagnosing, and monitoring patients with hematological disorders. High speed and broad applicability of flow cytometry allows for the diagnosis. Currently, there are no consensus panels being used; consequently, the leukemia & lymphoma (L&L) testing remains a single-vial antibody being used, with various in-house laboratory developed tests (LDTs) being used to test patient specimens. Furthermore, the analysis of flow cytometer generated data is not standardized and requires a high level of expertise and training for interpretation of complex data. Therefore, optimized and standardized immunostaining protocols for the diagnosis, classification, and prognostic sub-classification of hematological malignancies are needed.

Enrollment will occur at up to 8 investigational sites . Data will be acquired from Eligible remnant/leftover specimens on the BD FACSLyric flow cytometer and evaluated by site personnel and expert analysts .

The final diagnosis and the affected cell population will be determined by site standard of care .

Analysis of data will evaluate identification of 1) normal vs abnormal cell populations and 2) BCP-ALL, AML, and less certain diseases by the expert & site analysts as compared to the final diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Specimen collected/handled prior to enrollment in accordance with site policies and procedures.
2. Specimen with adequate volume (1 mL) to complete protocol tests.
3. Specimen is leftover PB and BM from routine flow cytometry laboratory testing for having or suspected of having acute leukemia disorders (i.e. AML, BCP-ALL, ALAL, etc.), myelodysplastic syndrome (MDS), other hematological, or non-hematological disorders.
4. Specimen from newly diagnosed or relapsed subject.
5. Only one specimen type (PB or BM) shall be enrolled per given subject.
6. Specimen is stored at room temperature, upon receipt by the site.
7. Specimens are collected in EDTA (K2 or K3) or heparin (sodium or lithium).
8. Age of specimen (BCP ALL T1: time of collection to start of first pre-wash; ALOT, AML T1-T4: time of collection to start of staining): ≤ 24 hours.
9. Specimens are from subjects irrespective of race, gender, and ethnicity

Exclusion Criteria:

1. Specimen is from healthy subject.
2. Specimen from subject <3 years of age.
3. Specimen is from subject undergoing any treatment for any form of leukemia.
4. Specimen is from subject with minimal residual disease (MRD) as determined by the site.
5. Specimen is from subject suspected of plasma cell disorders.
6. Visibly clotted specimen.
7. Visibly hemolyzed specimen.
8. Frozen specimen.
9. Refrigerated specimen.
10. Fixed specimen.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A minimum of evaluable 200 remnant/leftover peripheral blood and bone marrow specimens from routine flow cytometry laboratory testing for specimens from subjects 3 Years and older having or suspected of having acute leukemia disorders , myelodysplastic syndrome (MDS), and other hematological or non-hematological disorders. Specimens from healthy subjects will be excluded.
  At least 100 specimens must have abnormal lymphoid or myeloid cells, at least 100 must have normal lymphoid and myeloid cells.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Comparison between expert analysts' determination of normal and abnormal specimen and final diagnosis (Sensitivity Analysis) | Within 24 Hours of specimen collection
  Determine equivalence between the investigational OneFlow Acute Leukemia Panel on the BD FACSLyric system results analyzed by two independent experts versus the final clinical diagnosis for Normal (lymphoid and myeloid) or Abnormal (neoplastic lymphoid or myeloid) phenotypes.
  Sensitivity will be calculated
Comparison between expert analysts' determination of normal and abnormal specimen and final diagnosis (Specificity Analysis) | Within 24 Hours of specimen collection
  Determine equivalence between the investigational OneFlow Acute Leukemia Panel on the BD FACSLyric system results analyzed by two independent experts versus the final clinical diagnosis for Normal (lymphoid and myeloid) or Abnormal (neoplastic lymphoid or myeloid) phenotypes.
  Specificity will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Imelda Omana-Zapata, MD, PHD, Study Director — Becton, Dickinson and Company
Locations (8):
- United States (4):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - New York-Presbyterian Hospital Weill Cornell Medicine, New York, New York
  - University Of North Carolina, Chapel Hill, North Carolina
  - CorePath Laboratories, San Antonio, Texas
- Fleury Group, São Paulo, Brazil
- Motol University Hospital, Childhood Leukemia Investigation, Prague, Czechia
- University of Salamanca, Salamanca, Spain
- Cambridge University, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No